CLINICAL TRIAL: NCT05315895
Title: A Multi-Center Prospective Cohort Study of Dampness Syndrome in China
Brief Title: The Dampness Syndrome of Chinese Medicine Cohort Study
Acronym: DACOS
Status: Recruiting | Type: Observational
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: State Key Laboratory of Dampness Syndrome of Chinese Medicine, the Second Affiliated Hospital of Guangzhou University of Chinese Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: SZ2021ZZ06
Record Dates: First submitted 2022-03-11; First posted 2022-04-07 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Chronic Disease; Cancer; Dementia Alzheimers; Metabolic Disease; Aging; Alzheimer Disease, Early Onset
Keywords: Dampness Syndrome; multi-center study; prospective cohort study
MeSH Terms: conditions — Chronic Disease; Neoplasms; Alzheimer Disease; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — All biological specimens (including blood, feces, urine, saliva and tongue coating) will be stored in the biological resource center of the our research centers after written informed consent obtained from all subjects who voluntarily participated in this clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- general population: general population in a specific area and specifc time range.
  Interventions: Other: natural aging process

INTERVENTIONS:
Other: natural aging process — To observe the relationship between new cases of diseases and health status of people exposed to different factors such as life style, alcohol consumption, eating habits, etc.

SUMMARY:
The researchers plain to build a large-scale, longitudinal, prospective cohort characterized by TCM dampness syndrome. With the biobank of this cohort the investigators want to find the causality between TCM dampness syndrome and clinical chronic diseases and a new way to treat clinical disease.

DETAILED DESCRIPTION:
DACOS is a national large- scale, longitudinal, multi-center, prospective, cohort study of natural person aged 35 to 75. The baseline survey and the follow-up surveys will be conducted in 5 areas covering the eastern, northern, western, southern and middle parts of China. In this study 100,000 natural person will be regularly followed up for 5 years(visited once a year), with the loss rate ≤15%. Three parts will be carried in the form of interview, physical examination and biological sample collection. During the interview, the investigators plan to do some questionnaires to learn participants' demographic characteristics, life style, disease history, healthy condition(EQ-5D-5L, SDS,), cognition state(AD-8, MMSE, MoCA) and the results of TCM syndrome differentiation(Score of Dampness syndrome and TCM constitution scale). All biological specimens (including blood, feces, urine, saliva and tongue coating) will be collected and stored in the biological resource center until researchers request their use. With the building up of this cohort, the researchers will analyze the causality between dampness syndrome and specific chronic diseases such as diabetes, coronary heart disease, cancer, dementia and so on.

ELIGIBILITY:
Inclusion Criteria:

1. Residents aged 30 to 79, whose residence is consistent with their registered permanent residence location;
2. Residents who voluntarily participate in the project, agree to the collection of their biological information, and sign the informed consent form;
3. Residents who have no mental illness and other related diseases, and display a normal ability of expression and understanding;

Exclusion Criteria:

1. Residents who reject collaboration;
2. Residents who allow no follow-up visits.

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: general population in a specific area and specifc time range. Such as civil servants of Guangdong Province. Medical workers in Xinjiang.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
emerging diseases | through study completion, an average of 1 year
  This study will pay attention to the emerging situation of clinical chronic diseases, such as cancer, diabetes, hypertension, coronary heart disease, dementia, etc. Each follow-up the researchers will record the incidence of the emerging diseases of interviewees' by questionnaire including the name of the disease, time of onset and treatments.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment(MoCA) | through study completion, an average of 1 year
  MoCA is a brief, 30-question test that helps healthcare professionals detect cognitive impairments very early on, allowing for faster diagnosis and patient care. MoCA is the most sensitive test available for detecting Alzheimer's disease, measuring executive functions and multiple cognitive domains. The value range 0-30: higher scores mean a better Cognitine. The score above 26 is considered the normal congnitive level
European Quality of Life 5-dimensional questionnaire (EQ-5D-5L) | through study completion, an average of 1 year
  The EQ-5D comprises five dimensions of health: mobility, ability to self-care, ability to undertake usual activities, pain and discomfort, and anxiety and depression. . EQ-5D-5L, includes five levels of severity for each dimension (no problems, slight problems, moderate problems, severe problems, and extreme problems). The value range 0-100: higher scores mean a worse outcome.
Mini-Mental State Exam (MMSE) | through study completion, an average of 1 year
  MMSE is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills. The value range 0-30: higher scores mean a better Cognitine.
interview questionnaire | through study completion, an average of 1 year
  Demographic characteristic, life style. disease history, allergies will be involoved.
change of the blood routine results | through study completion, an average of 1 year
  WBC, RBC, PLT , HB, NEUT% and LYM% will be tested and recorded. Above or below each mormal value will be considered as abnormal.
urine routine | through study completion, an average of 1 year
  urinary WBC and urinary RBC will be observed. negative or below 5/HP is normal.
  BLO and GLU and PRO in urine will also be test. Negative is normal.
change of faeces routine | through study completion, an average of 1 year
  cells in faeces will be tested such as RBC and WBC. Negative occult blood（FOB) is difined normal.
change of hepatic function | an average of 1 year
  The researchers will check the results of ALT and AST. TBil, DBIL, TBA and TP, ALB. Any indices above or below the criteria range is defined as abnormal. Every time point investigators will record the change of these indices.
change of renal function | an average of 1 year
  The researchers will check the results of Cr， BUN, TC， LDL， HDL,UA and fasting blood glucose，glycosylanted. Any indices above or below the criteria range is defined as abnormal. Every time point investigators will record the change of these indices.
change of CRP | an average of 1 year
  change of CPP
change of Hcy | an average of 1 year
  change of Hcy
change of thyroid function | an average of 1 year
  change of TSH ,FT3, FT4
change of Vit B12 and folic acid | an average of 1 year
  change of Vit B12
change of coagulation function | an average of 1 year
  change of PT, INR,TT,APTT，FIB
change of abdominal ultrasound | an average of 1 year
  change of abdominal ultrasound
change of gynecologic ultrasound | an average of 1 year
  change of gynecologic ultrasound
change of ECG | an average of 1 year
  The researchers will check the change of P, QRS and ST segments separately in electrocardiogram.
change of brain MRI | an average of 1 year
  change of brain MRI. The investigators will focus on the change of hippocampal volume and the spacing of temporal sulcus gyrus.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Province Hospital of Tradtional Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
If you need to access or use the population information database and biological sample database, you must go through strict application and approval processes at first
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After half year of the baseline and follow-ups data completing.
Access Criteria: A professional qualification panel determines whether the visitor is qualified to view and use the repository.

REFERENCES:
- [Derived] Li M, Liu N, Jiang G, Zeng H, Guo J, Wu D, Zhou H, Wen Z, Zhou L. Health-related quality of life in populations with diabetes, prediabetes, and normal glycemic levels in Guangzhou, China: a cross-sectional study. Front Endocrinol (Lausanne). 2025 May 23;16:1518204. doi: 10.3389/fendo.2025.1518204. eCollection 2025. PMID 40487765